CLINICAL TRIAL: NCT00929409
Title: A 6-week Randomised, Open Comparative, Multi-centre Study of Intravenous Ferric Carboxymaltose (Ferinject) and Oral Iron (Duroferon) for Treatment of Post Partum Anemia
Brief Title: Controlled Randomised Trial of Ferric Carboxymaltose and Oral Iron to Treat Postpartum Anemia
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Stopped prematurely because too few patients were recruited.
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Sykehuset Innlandet HF (Other); Sykehuset Buskerud HF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4.2009.373; 21830 (Other: NSD, Norway); 09/03045-4 (Other: SLV, Norway); 2008-008526-79 (EudraCT Number)
Record Dates: First submitted 2009-06-26; First posted 2009-06-29 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Anemia, Iron-Deficiency; Puerperal Disorders; Depression, Postpartum
Keywords: Postpartum anemia, iron-deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency; Puerperal Disorders; Depression, Postpartum | interventions — ferric carboxymaltose; Iron-Dextran Complex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peroral iron - ferrous sulfate tablets (Active Comparator): Peroral iron given as one tablet of ferrous sulfate 100 mg two times daily
  Interventions: Drug: Ferrous sulfate tablets
- Ferric carboxymaltose (Active Comparator): Intravenous infusion of Ferric Carboxymaltose (Ferinject), the given dose is adapted according to the individual patient's requirement. No other form of iron supplementation is given.
  Interventions: Drug: Ferric carboxymaltose

INTERVENTIONS:
Drug: Ferric carboxymaltose — Intravenous infusion of Ferric carboxymaltose in a dose calculated to meet the individual patient's requirements following the Ganzoni formula
  Other Names: Ferinject
  Arms: Ferric carboxymaltose
Drug: Ferrous sulfate tablets — Standard tablets containing 100 mg ferrous sulfate, 1 tablet two times daily
  Other Names: Duroferon
  Arms: Peroral iron - ferrous sulfate tablets

SUMMARY:
200 patients with post partum anemia will be randomised to receive either intravenous iron (intervention group) or peroral iron (control group).

The hypothesis is that intravenous iron supplementation is superior to standard peroral iron.

DETAILED DESCRIPTION:
The study is a multi center phase 3 trial, comprising 3 medium sized obstetrical units in Norway.

The amount of iron given to the intervention group is calculated according to the modified Ganzoni formula. The control group is given the standard regime of 200 mg ferro sulphate daily. In both groups, treatment start at inclusion, within 48 h of delivery.

The sample size was based on power calculations: About 200 participants are required to detect a difference of 0.5 g/dl between the groups (with 80 % power).

Randomization is performed by use of opaque envelopes. An electronic CRF is applied. Laboratory analysis are provided by a recognized Swedish biochemical laboratory.

Apart from hemoglobin and the common iron parameters, the serum concentration of soluble ferritin receptors will be analyzed, as well as hepcidin levels.

ELIGIBILITY:
Inclusion Criteria:

* Woman within 48 h post partum
* Hemoglobin level equal or higher than 6.5 g/dl and equal or lower than 8.5 g/dl
* Able to read and understand the Norwegian language
* Signed informed consent

Exclusion Criteria:

* Anemia not attributable to iron deficiency
* Contraindications for any of the study drugs
* Treatment with drugs, dietary supplements or natural remedies containing iron
* Clinically significant condition which in the opinion of the investigator should disqualify the patient from the study
* Assessed as requiring blood transfusion(s)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Haemoglobin concentration | 6 weeks

SECONDARY OUTCOMES:
Ferritin | 6 weeks
Fatigue | 6 weeks
  Fatigue scale
Quality of life | 6 weeks
  SF-36
Post partum depression | 6 weeks
  Edinburgh Post Partum Depression Scale

CONTACTS AND LOCATIONS:
Overall Officials: Bjorn Backe, MD PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (3):
- Norway (3):
  - Department of Obstetrics, Vestre Viken Hospital Trust, Drammen
  - Sykehuset Innlandet HF, Lillehammer
  - St Olavs Hospital, Trondheim